CLINICAL TRIAL: NCT00212784
Title: A Phase III, Double-Blind, Randomized, Active-Controlled, Two-Armed, Multicenter, Efficacy and Safety Assessment (ACTAMESA) of Org 5222 and Olanzapine in the Treatment of Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Efficacy and Safety of Asenapine Using an Active Control in Subjects With Schizophrenia or Schizoaffective Disorder (25517)(P05935)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05935; ACTAMESA, 25517
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: asenapine
- Arm 2 (Active Comparator)
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: asenapine — Flexible dose, 1-2 tablets sublingual two times per day (1 or 2 tablets in the morning and 1 or 2 tablets in the evening). Each tablet contains either 5 mg asenapine or matching placebo.
  Other Names: Org 5222; SCH 900274
  Arms: Arm 1
Drug: olanzapine — Oral capsules (5 mg or placebo); 1 to 2 tablets twice daily
  Arms: Arm 2

SUMMARY:
The primary features of schizophrenia and schizoaffective disorder are characterized by positive (inability to think clearly and distinguish reality from fantasy) and negative symptoms (reduction or absence of normal behavior or emotions). Other symptoms include reduced ability to recall and learn information, difficulty in problem solving or maintaining productive employment. Asenapine is an investigational drug that may help to correct the above characteristics of schizophrenia by altering the inbalance of brain hormones such as dopamine and serotonin. This is a 12-month trial that will test the efficacy and safety of asenapine using an active comparator (olanzapine) in the treatment of patients with schizophrenia. Patients who complete the 12-month trial will have the option of continuing on drug until the treatment code for the 12-month trial is unblinded.

ELIGIBILITY:
Inclusion Criteria:

* Subject with schizophrenia or schizoaffective disorder. Subject must sign a written informed consent.

Exclusion Criteria:

* Have an uncontrolled, unstable, clinically significant medical condition. Have any other psychiatric disorder other than schizophrenia as a primary diagnosis including depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1225 (Actual)
Dates: Start 2003-09-04 (Actual); Primary Completion 2006-03-15 (Actual); Study Completion 2006-03-15 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS score at endpoint (52-week double-blind or last assessment after baseline) from baseline | Screening, Baseline, Week 2, 4, 6, 8, 12, 20, 28, 36, 44, 52 (endpoint)

SECONDARY OUTCOMES:
Changes in PANSS subscale scores and Marder factor scores | At weeks 2, 4, 6, 8, 12, 20, 28, 36, 44 and endpoint
Changes in CGI-S | At each assessment time point from baseline
Patient functionality and subjective well-being (as measured by LOF, SF-12 and SWN) | At weeks 8, 20, 28, 36, 44 and endpoint
Severity of depressed mood (as measured by the Calgary Depression Scale for Schizophrenia) | At weeks 6, 28 and endpoint
Resource utilization (as measured by frequency and length of hospital stay) | During the study period
Satisfaction with treatment in comparison with previous treatment as assessed by the investigator and patient) | At endpoint
Population kinetics | Plasma samples at weeks 2 and 6 in comparison with baseline
Pharmacogenetics (as part of a global effort to investigate possible associations between genetic polymorphisms in relation to response to asenapine and related drugs and in relation to characteristics of schizophrenia and related conditions) | During the study period
Safety and tolerability: EPS (AIMS, BARS, SARS) | At weeks 1, 3, 6, 16, 24, 32, 40 and endpoint
Adverse Events | continuously and up to 7 days after endpoint
Pregnancy Test | At endpoint
Blood Test | At weeks 1, 3, 6, 16, 24, 32, 40 and endpoint
Weight and vital signs | at all assessment time points from baseline
ECGs | Weeks 3, 6, 24, and endpoint

REFERENCES:
- [Result] Schoemaker J, Naber D, Vrijland P, Panagides J, Emsley R. Long-term assessment of Asenapine vs. Olanzapine in patients with schizophrenia or schizoaffective disorder. Pharmacopsychiatry. 2010 Jun;43(4):138-46. doi: 10.1055/s-0030-1248313. Epub 2010 Mar 4. PMID 20205074